CLINICAL TRIAL: NCT03572842
Title: Functional Non Specific Immunity Monitoring After Kidney Transplantation Using an Interferon Gamma Test, QuantiFERON Monitor®
Brief Title: Functional Non Specific Immunity Monitoring After Kidney Transplantation Using an Interferon Gamma Test
Acronym: QuantiFERON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-AOI-04
Record Dates: First submitted 2018-05-29; First posted 2018-06-28 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- quantiferon monitor (Other): Test measuring interferon gamma production after T cells and Natural Killers (NK) in vitro stimulation : QuantiFERON Monitor® (QFM)
  Interventions: Other: quantiferon monitor test

INTERVENTIONS:
Other: quantiferon monitor test — different blood test with quantiferon monitor

SUMMARY:
The best renal replacement therapy is kidney transplantation. It improves end-stage renal kidney disease (ESRD) patients quality of life and increases their survival, but still remains risky. Morbidity in kidney transplantation is dominated by two main complications : acute graft rejection and infections. To maintain an accurate balance between rejection and infection, immunosuppressive therapy must to be used with caution and kept into a tight spectrum.

The investigators dispose of a new test measuring interferon gamma production after T cells and Natural Killers (NK) in vitro stimulation : QuantiFERON Monitor® (QFM). They hypothesized QFM monitoring could improve management after kidney transplantation providing functional immune data to optimize balance between rejection and infection.

The investigators aim to assess whether QFM could be an objective biomarker to predict infection and rejection risks after kidney transplantation.

DETAILED DESCRIPTION:
The best renal replacement therapy is kidney transplantation. It improves end-stage renal kidney disease (ESRD) patients quality of life and increases their survival, but still remains risky. Morbidity in kidney transplantation is dominated by two main complications : acute graft rejection and infections. According to literature, acute rejection appears in more than 10% of kidney graft recipients. The first month after transplantation is frequently affected by bacterial infections such as pneumopathies (4.5 to 16%), urinary tract infections (22.7 to 56.7 %), surgical site infections (7.3 to 18.5%) and bacteremia (3.5 to 4.6%). Then, during the first year, infections, most of them opportunist ones, are essentially due to cytomegalovirus (8%), BK virus (most than 10%) and herpes simplex reactivation (most than 50%). Those immunosuppressed patients can also develop community acquired infections : respiratory tract infections (flu or bacterial pneumonias) or urinary tract infections. Therefore, long-term anticalcineurin use can lead to chronic graft dysfunction. To maintain an accurate balance between rejection and infection, immunosuppressive therapy must to be used with caution and kept into a tight spectrum. To guide physicians maintaining this balance, therapeutic drug monitoring is performed in routine.

An objective marker for cellular immune response, based on cellular immunodeficiency status specific for each patient could, guide a personalized immunosuppressive treatment. The investigators now dispose of a new test measuring interferon gamma production after T cells and Natural Killers (NK) in vitro stimulation : QuantiFERON Monitor® (QFM). They hypothesized QFM monitoring could improve management after kidney transplantation providing functional immune data to optimize balance between rejection and infection.

The best renal replacement therapy is kidney transplantation. It improves end-stage renal kidney disease (ESRD) patients quality of life and increases their survival, but still remains risky. Morbidity in kidney transplantation is dominated by two main complications : acute graft rejection and infections. According to literature, acute rejection appears in more than 10% of kidney graft recipients. The first month after transplantation is frequently affected by bacterial infections such as pneumopathies (4.5 to 16%), urinary tract infections (22.7 to 56.7 %), surgical site infections (7.3 to 18.5%) and bacteremia (3.5 to 4.6%). Then, during the first year, infections, most of them opportunist ones, are essentially due to cytomegalovirus (8%), BK virus (most than 10%) and herpes simplex reactivation (most than 50%). Those immunosuppressed patients can also develop community acquired infections : respiratory tract infections (flu or bacterial pneumonias) or urinary tract infections. Therefore, long-term anticalcineurin use can lead to chronic graft dysfunction. To maintain an accurate balance between rejection and infection, immunosuppressive therapy must to be used with caution and kept into a tight spectrum. To guide physicians maintaining this balance, therapeutic drug monitoring is performed in routine.

An objective marker for cellular immune response, based on cellular immunodeficiency status specific for each patient could, guide a personalized immunosuppressive treatment. The investigators now dispose of a new test measuring interferon gamma production after T cells and Natural Killers (NK) in vitro stimulation : QuantiFERON Monitor® (QFM). They hypothesized QFM monitoring could improve management after kidney transplantation providing functional immune data to optimize balance between rejection and infection.

They aim to assess whether QFM could be an objective biomarker to predict infection and rejection risks after kidney transplantation.

The investigators plan to perform a monocentric interventional prospective study. They will dose QFM at D0, before patients discharge (between D7 and D21), M3 and M6 after kidney transplantation. Patients will be followed up to 24 months.

Their primary endpoint will be non specific cellular immunity evaluation after kidney transplantation using serial measurements of QFM. Their secondary endpoints will be : (i) correlate QFM levels with infectious risk, (ii) and with graft rejection, (iii) correlate QFM levels with lymphocytes sub-populations monitoring.

The investigators aim to assess whether QFM could be an objective biomarker to predict infection and rejection risks after kidney transplantation.

They plan to perform a monocentric interventional prospective study. They will dose QFM at D0, before patients discharge (between D7 and D21), M3 and M6 after kidney transplantation. Patients will be followed up to 24 months. Their primary endpoint will be non specific cellular immunity evaluation after kidney transplantation using serial measurements of QFM. The investigator's secondary endpoints will be : (i) correlate QFM levels with infectious risk, (ii) and with graft rejection, (iii) correlate QFM levels with lymphocytes sub-populations monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation in Nice University Hospital during the inclusion period
* Free and informed consent
* Age > 18 years-old

Exclusion Criteria:

* Current infection
* Vulnerable people (minors, guardianship or curatorship, pregnant women, deprivation of liberty, person who does not speak French)
* Non-affiliated person with Social Security
* Kidney transplantation contraindication Exclusion criterion
* Transplantectomy before sixth month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Change of QuantiFERON Monitor® levels (interferon gamma, UI/mL) | At day 0 (inclusion), Between Day 7 and Day 21 (before discharge), 3 month post-transplantation, 6 month post-transplantation
  QuantiFERON Monitor® levels (interferon gamma, UI/mL)

SECONDARY OUTCOMES:
Acute cellular and/or antibodies mediated graft rejection | At day 0 (inclusion), Between Day 7 and Day 21 (before discharge), 3 month post-transplantation, 6 month post-transplantation
  Acute cellular and/or antibodies mediated graft rejection
Infections | At day 0 (inclusion), Between Day 7 and Day 21 (before discharge), 3 month post-transplantation, 6 month post-transplantation
  occurence of infections
Lymphocytes sub-populations | At day 0 (inclusion), Between Day 7 and Day 21 (before discharge), 3 month post-transplantation, 6 month post-transplantation
  Lymphocytes sub-populations

CONTACTS AND LOCATIONS:
Overall Officials: Barbara SEITZ-POLSKI, Dr, Study Chair — Nephrology Department, Nice University Hospital; Marion CREMONI GAUCI, Principal Investigator — Nephrology Department, Nice University Hospital
Locations (1):
- Nephrology Department, Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No